CLINICAL TRIAL: NCT03025854
Title: Prospective Study for Prognostic Biomarkers of Nasopharyngeal Carcinoma
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Collaborators: Guilin Medical University, China (Other); First People's Hospital of Foshan (Other)
Responsible Party: Principal Investigator, Jun Ma, MD, Prof, Sun Yat-sen University
Other Study IDs: 2016-FXY-058
Record Dates: First submitted 2017-01-18; First posted 2017-01-20 (Estimated); Last update posted 2020-10-12 (Actual); Status verified 2020-10

CONDITIONS: Nasopharyngeal Carcinoma
MeSH Terms: conditions — Nasopharyngeal Carcinoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood and tumor tissue
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The purpose of this clinical research project is to explore potential biomarkers and validate the predictive and prognostic value of molecular signature in nasopharyngeal carcinoma.

DETAILED DESCRIPTION:
Objectives:

Primary: Evaluation of failure-free survival after three years of patients of nasopharyngeal carcinoma.

Secondary: Evaluation of overall survival after three years of patients of nasopharyngeal carcinoma.

Outline: This is a multicenter observational study. Tumor tissue specimens are obtained from the Sun Yat-sen University Cancer Center and Affiliated Hospital of Guilin Medical University. The samples are analyzed for biomarkers. The biomarkers are correlated with clinical outcomes (failure-free survival, overall survival, tumor response to treatment, distant metastasis, recurrence and death).

The aim of the analysis is to explore potential biomarkers and validate the predictive and prognostic value of molecular signature in nasopharyngeal carcinoma. This will lead to the definition of risk groups and stratification of patients and will help to precision medicine of nasopharyngeal carcinoma.

ELIGIBILITY:
Inclusion Criteria:

* Patients with newly histologically confirmed nasopharyngeal carcinoma
* No evidence of distant metastasis (M0)
* Written informed consent

Exclusion Criteria:

* Treatment with palliative intent

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with newly histologically confirmed nasopharyngeal carcinoma and no evidence of distant metastasis
Sampling Method: Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2017-01 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2023-01 (Estimated)

PRIMARY OUTCOMES:
Failure-free Survival | 3 years

SECONDARY OUTCOMES:
Overall Survival | 3 years

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided